CLINICAL TRIAL: NCT02102035
Title: Direct and Reversed Dorsal Digital Island Flaps: A Review of 65 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TSChen8992
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-10

CONDITIONS: Soft Tissue Reconstruction; Sensory Restoration
Keywords: defect; dorsal branch of the proper digital nerve; dorsal digital island flap; sensory reconstruction.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dorsal digital island flap (Other): The flap is used to cover the soft-tissue defects of the fingers.
  Interventions: Procedure: Direct and reversed dorsal digital island flap

INTERVENTIONS:
Procedure: Direct and reversed dorsal digital island flap — The direct dorsal digital island flap is used to cover the defects of adjacent fingers. The reversed dorsal digital island flap is used to cover the defects of the same fingers.

SUMMARY:
Reconstruction of soft tissue defects in the fingers continues to be a challenge problem. The study reports reconstruction of small to moderate defects of the fingers with the direct and reversed dorsal digital island flaps and evaluates the results of the use of the flaps.The main outcomes are static 2-point discrimination and Semmes-Weinstein monofilament scores of the flap and joint motion.

DETAILED DESCRIPTION:
At final follow-up, sensory restoration of the flap is measured using the static 2-point discrimination (2PD) test and Semmes-Weinstein monofilament (SWM) test. Active motion of the joints is measured using a standard hand goniometer. For the direct DDIF, total active motion is calculated as the sum of degrees of active flexion of the interphalangeal and the metacarpophalangeal joints subtracted from the degrees of extension deficit. For the reversed DDIF, total active motion of the donor finger is calculated as the sum of degrees of active flexion of the proximal and distal interphalangeal joints subtracted from the degrees of extension deficit.

ELIGIBILITY:
Inclusion Criteria:

* a defect greater than or equal to 1.5 cm in length
* the defects on the dorsal and lateral aspects of the fingers
* the defects located between the distal 1/2 of the middle phalanx and the tip of the finger
* a patient between 15 and 60 years of age.

Exclusion Criteria:

* injuries involving the donor sites or the course of the vascular pedicle
* a defect less than 1.5 cm in length.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Static 2-point discrimination test | 16 to 24 months
  The test points are at the center of the flap. Each area is tested 3 times with a Discriminator (Ali Med, Dedham, MA). We stop at 4mm as a limit of static 2-point discrimination test and consider this normal.

SECONDARY OUTCOMES:
Total active motion | 16-24 months
  Active motion of the joints is measured using a standard hand goniometer. For the direct DDIF, total active motion is calculated as the sum of degrees of active flexion of the interphalangeal and the metacarpophalangeal joints subtracted from the degrees of extension deficit. For the reversed DDIF, TAM of the donor finger is calculated as the sum of degrees of active flexion of the proximal and distal interphalangeal joints subtracted from the degrees of extension deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Tang P, Zhang L. Reconstruction of a soft tissue defect in the finger using the heterodigital neurocutaneous island flap. Injury. 2013 Nov;44(11):1607-14. doi: 10.1016/j.injury.2013.06.025. Epub 2013 Jul 18. PMID 23871427